CLINICAL TRIAL: NCT07041814
Title: Bayesian Pragmatic Trial for Pubertal Induction in Turner Syndrome: TRansformation Initiative For Efficient Clinical TriAl Design Advancement in RarE Diseases (TRIFECTA-DARED Framework)
Brief Title: A Study Comparing Different Treatment Approaches for the Initiation of Puberty in Girls With Turner Syndrome Using a TRIFECTA-DARED Approach for Rare Diseases
Acronym: TRIFECTA-DARED
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUP-2024-011; NMRR ID-25-02169-7TA (Registry Identifier: National Medical Research Registry (Malaysia))
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Turner Syndrome
Keywords: Turner Syndrome; Hormone Replacement Therapy; Progynova; Oestrogel; Transdermal 17β Estradiol; Estradiol Valerate; Pubertal Induction
MeSH Terms: conditions — Turner Syndrome | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Estradiol Valerate (Progynova) (Active Comparator): Progynova is an oral hormone replacement therapy containing the active ingredient estradiol valerate, a synthetic ester of 17β-estradiol that, upon ingestion, is rapidly converted to bioidentical estradiol. Each film-coated tablet delivers either 1 mg or 2 mg of estradiol valerate, with inactive excipients including lactose monohydrate, maize starch, povidone, magnesium stearate, and hypromellose. Progynova tablets are supplied in blister packs of 28 tablets, with recommended storage at room temperature (15-30 °C), protected from moisture and direct sunlight. In this trial, Progynova will be administered starting at 1 mg twice weekly and titrated up to 4 mg daily over an 18-month period, in accordance with local clinical guidelines for pubertal induction in Turner Syndrome.
  Interventions: Drug: Oral estradiol valerate
- Transdermal 17β estradiol (Oestrogel®) (Experimental): Oestrogel® is a transdermal hormone replacement therapy containing 17β-estradiol in a hydroalcoholic gel formulation designed for topical application. Each pump actuation delivers 0.75 mg of estradiol in a 1.25 g dose of gel, which is formulated with excipients including ethanol, propylene glycol, carbomer, sodium hydroxide, and purified water to ensure consistent hormone release and skin penetration. The gel is supplied in multi-dose pump bottles (150 g), each providing up to 120 actuations. In this trial, Oestrogel® will be administered starting at one pump actuation (0.75 mg) twice weekly, with dose escalation every 3 months according to predefined protocol milestones, up to a maximum of four actuations daily (3 mg estradiol) over an 18-month induction period. Participants will be instructed on correct application technique-applying gel to clean, dry skin and allowing at least 5 minutes for drying before dressing-to ensure optimal absorption and minimize residue transfer
  Interventions: Drug: Transdermal 17β estradiol

INTERVENTIONS:
Drug: Oral estradiol valerate — Progynova is an oral hormone replacement therapy containing the active ingredient estradiol valerate, a synthetic ester of 17β-estradiol that, upon ingestion, is rapidly converted to bioidentical estradiol. Each film-coated tablet delivers either 1 mg or 2 mg of estradiol valerate, with inactive excipients including lactose monohydrate, maize starch, povidone, magnesium stearate, and hypromellose. In terms of pharmacokinetics, oral estradiol valerate undergoes first-pass metabolism in the liver, yielding a peak serum estradiol concentration within 4-8 hours of dosing and a biological half-life of approximately 20 hours. Progynova tablets are supplied in blister packs of 28 tablets, with recommended storage at room temperature (15-30 °C), protected from moisture and direct sunlight.
  Arms: Oral Estradiol Valerate (Progynova)
Drug: Transdermal 17β estradiol — Oestrogel® is a transdermal hormone replacement therapy containing 17β-estradiol in a hydroalcoholic gel formulation designed for topical application. Each pump actuation delivers 0.75 mg of estradiol in a 1.25 g dose of gel, which is formulated with excipients including ethanol, propylene glycol, carbomer, sodium hydroxide, and purified water to ensure consistent hormone release and skin penetration. Upon application to intact skin-typically the forearm or thigh-the gel allows for direct systemic absorption of estradiol, bypassing first-pass hepatic metabolism. Peak serum estradiol levels are generally reached within 6-12 hours post-application, with a half-life of approximately 10-20 hours, resulting in more physiological, steady- steady-state estradiol exposure compared to oral formulations. The gel is supplied in multi-dose pump bottles (150 g), each providing up to 120 actuations.
  Arms: Transdermal 17β estradiol (Oestrogel®)

SUMMARY:
Turner syndrome is a condition in which a girl's body does not make enough estrogen on its own, so doctors give estrogen to help start breast and uterine (womb) development. Hence, the goal of this clinical trial is to learn whether two different ways of giving estrogen help girls and young women with Turner syndrome go through puberty normally, and to compare how well each method works and how safe they are.

The main questions the trial aims to answer are:

1. Does taking an oral estrogen tablet (Progynova) or applying an estrogen gel (Oestrogel) lead to better breast development?
2. Does one method lead to a larger uterine size as seen on ultrasound?
3. Do participants start menstrual-like (withdrawal) bleeding, and does one method cause it sooner?
4. What side effects (for example, headaches, nausea, changes in blood tests) happen with each method?

Who can take part?

* Girls and young women aged 11-30 years with a confirmed diagnosis of Turner syndrome and no previous estrogen treatment.
* They have not yet begun puberty (no breast growth, and a small uterus on ultrasound).
* They agree to adhere to the study schedule and keep a diary of any bleeding or side effects

What will happen to the participants during the clinical trial?

* Get assigned at random to one of two groups (1:1 ratio):

  1. Gel group: Apply Oestrogel (17β-estradiol) to the skin, starting twice a week, then daily with increasing doses over 19 months.
  2. Tablet group: Swallow Progynova (estradiol valerate) tablets, starting twice a week, then daily with increasing doses over 19 months.
* Visit the clinic at the start of study (baseline), month 1, 7, 13, and 19 for:

  1. A physical exam (including breast staging).
  2. An ultrasound to measure uterine length and thickness.
  3. A blood test for safety checks (triglycerides and other markers).
  4. Keep a diary noting any spotting or bleeding (called withdrawal bleeding) and any side effects.

Why does this matter?

Girls and young women with Turner syndrome often need estrogen to begin puberty safely. This trial will show which method-gel or tablets-best mimics natural puberty (breast and uterine growth), how quickly menstrual-like bleeding begins, and which has fewer unwanted effects. The findings will help doctors choose the most effective and safe treatment for people with Turner syndrome.

DETAILED DESCRIPTION:
Turner syndrome (TS) is a chromosomal condition in which the loss of one X chromosome leads to ovarian failure, absent or delayed natural puberty, reduced bone density, and elevated cardiovascular and metabolic risk. This interventional, Bayesian Phase II pragmatic trial is being undertaken within the TRIFECTA-DARED framework to address a critical gap in the management of pubertal induction for adolescent and young adult females with TS. While estrogen replacement therapies are standard, there remains uncertainty about which regimen best approximates natural pubertal development, optimizes uterine growth, and minimizes adverse metabolic or thromboembolic risks. Our trial arises from the need for robust, locally generated evidence in Malaysia to inform clinical practice in this rare-disease context.

This single-centre study, conducted at Hospital Canselor Tuanku Muhriz (HCTM) and Hospital Pakar Kanak-Kanak at the Cheras Campus of Universiti Kebangsaan Malaysia, received ethics approval from the Universiti Kebangsaan Malaysia Research Ethics Committee (UKMREC). The trial design uses an open-label, randomized,1:1 ratio design, augmented by matched historical control data. After providing informed consent, participants are allocated by a central, computer-generated sequence (stratified by age category and body mass index) to receive either oral estradiol valerate (Progynova) or transdermal 17β-estradiol gel (Oestrogel). Treating clinicians and participants remain unblinded, while the trial statistician is masked until the database lock.

Both regimens begin with twice-weekly dosing for the first four weeks, followed by once-daily administration for the remaining 18 months. Incremental dose doubling at month 7 and again at month 13 is designed to mimic the gradual rise in endogenous estradiol characteristic of normal puberty. Doses are dispensed and tracked through an electronic case report form (eCRF) with real-time logging of medication issuance and returns, and participants maintain a daily diary to record dosing adherence, any spotting or bleeding episodes, and all adverse experiences.

Scheduled study visits occur at baseline and at months 7, 13, and 19, with quarterly safety check-ins during the first year. At each visit, a pediatric or adolescent gynecologist performs a comprehensive physical examination-including growth measurements, vital signs, and breast development staging-and obtains a transabdominal ultrasound to document uterine dimensions. Blood samples are drawn for routine safety laboratories (liver function, lipid profile, complete blood count) and hormone assays.

Safety oversight is provided by an independent Data Monitoring Committee (DMC), which reviews periodic safety reports prepared by an external statistician. Adverse events are graded per the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Any life-threatening or disabling event associated with the study drug triggers immediate notification to the ethics committee and regulatory authorities within 24 hours; other Grade 3 or higher events are reported within five business days. Prespecified halting criteria include unexplained severe laboratory abnormalities, life-threatening reactions deemed drug-related, or anaphylactic-type responses within 24 hours of dosing.

All data are captured in a secure REDCap eCRF with built-in validation and audit trails. Concomitant medications are coded using the World Health Organization Anatomical Therapeutic Chemical (WHO-ATC ) classification system, and adverse events use MedDRA terminology. The database is backed up daily across multiple secure servers and locked after each monitoring visit. Quality assurance involves internal audits every six months by the sponsor, all in accordance with Good Clinical Practice (GCP) standards.

Data analysis follows an intention-to-treat framework with multiple imputation for missing values and sensitivity checks in a per-protocol subset. Although specific outcome measures are recorded elsewhere, continuous and categorical data will be analyzed using appropriate statistical models. In addition, Bayesian hierarchical modelling will be carried out to incorporate informative priors derived from matched historical TS cohorts, yielding posterior estimates of treatment effects and enabling predictive checks, thus providing robust inference despite the small sample inherent to this rare-disease study.

The trial is registered on ClinicalTrials.gov and the Malaysian National Medical Research Registry. Aggregate results will be posted within six months of study completion and disseminated through peer-reviewed publications and conference presentations following International Committee of Medical Journal Editors (ICMJE) authorship guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 11-30 years old with karyotype-verified (45, X or other similar karyotypes) and clinically confirmed Turner's syndrome prior at the time of pubertal induction
2. Confirmed estrogen deficiency with primary ovarian failure (high level of follicular stimulating hormone (FSH > 25 IU/L))
3. Patients who have not undergone pubertal development ( no breast development and underdeveloped uterus size).
4. Hormone Replacement Therapy (HRT)-naive TS patients
5. Breast Tanner Stage of 2 or less.
6. Patients on Growth Hormone (GH) will be allowed entry into the study.
7. Consented to trial participation (from individual TS patients (if aged 18 and above) or the parents or guardians (for under-18 TS patients) with individual's assent

Exclusion Criteria:

1. Patients with signs of spontaneous puberty
2. Contraindications to trial products (e.g hypersensitivity to any components of the HRT) based on the most recent version of the British National Formulary (BNF 85)
3. Previous history of exposure to estrogen treatment.
4. Concomitant use of other drugs that affect the bone mineral density (BMD) of the participants (e.g. Bisphosphonates or prolonged use of systemic corticosteroids). Vitamin D supplementation and short corticosteroid usage are allowed.
5. Acute or chronic hepatic disease
6. Patients with untreated hypothyroidism
7. Inflammatory bowel disease (Ulcerative Colitis, Crohn's disease) and coeliac disease
8. Cigarette-smoking patients
9. Severely obese patients based on the following criteria:

   1. For TS patients aged 11-17 years old: Based on the WHO chart with BMI > 95th percentile
   2. For TS patients aged 18 years until 30 years: BMI of 37.5 or above based on the Malaysian Clinical Practice Guideline for the Management of Obesity
10. Unknown abnormal genital bleeding
11. Porphyria
12. Recent involvement with clinical research studies (previous 6 months) investigating new HRT formulations

Ages: 11 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportions of Turner Syndrome with Satisfactory Breast Development (defined as Turner Breast Stage 3 (B3) and above) | From enrollment (baseline) to 19 months after the commencement of intervention (end of follow-up)
  Tanner Staging System for Breast Development as assessed by a trained pediatric and adolescent gynaecologist specialist at Hospital Canselor Tuanku Muhriz (HCTM)'s Pediatric and Adolescent Gynaecology (PAG) Unit. Tanner Staging System has a range between Tanner Breast Stage 1 (B1) (minimum value) and Tanner Breast Stage 5 (B5) (maximum value). Each stage is classified as follows:
  B1: Prepubertal - no glandular tissue. Only the nipple is raised. B2: Breast bud stage - small mound forms. Areola begins to enlarge. B3: Further enlargement of the breast and areola with no separation of their contours.
  B4: Areola and nipple form a secondary mound above the level of the breast. B5: Mature adult breast - breast contour is smooth. The areola recedes to the general contour of the breast (although in some women, the areola may remain raised).
  Higher Tanner breast stage means better breast development (i.e. better outcome)
Median time to achieving Tanner Breast Stage 4 (B4) and above (in days) | From enrollment to 19 months after the commencement of interventions (end of follow-up)
  Tanner Staging System for the assessment of Breast Development as assessed by the paediatric and adolescent gynaecology specialist at Hospital Canselor Tuanku Muhriz (HCTM)'s Pediatric and Adolescent Gynaecologist. Tanner Staging System has a range between Tanner Breast Stage 1 (B1) (minimum value) and Tanner Breast Stage 5 (B5) (maximum value). Each stage is classified as follows:
  B1: Prepubertal - no glandular tissue. Only the nipple is raised. B2: Breast bud stage - small mound forms. Areola begins to enlarge. B3: Further enlargement of the breast and areola with no separation of their contours.
  B4: Areola and nipple form a secondary mound above the level of the breast. B5: Mature adult breast - breast contour is smooth. Areola recedes to the general contour of the breast (although in some women areola may remain raised).
  Higher Tanner breast stage means better breast development (i.e. better outcome)
Uterine length (in cm) | From enrollment to 19 months after the commencement of interventions (end of follow-up)
  Ultrasonographic scan conducted at the Paediatric and Adolescent Gynaecology (PAG) unit performed by a trained PAG Specialist (trial outcome assessor)
Anteroposterior uterine fundal diameter (in cm) | From enrollment to 19 months after the commencement of intervention (end of follow-up)
  Ultrasonographic scan conducted at the Paediatric and Adolescent Gynaecology (PAG) unit, performed by a trained PAG Specialist (trial outcome assessor)

SECONDARY OUTCOMES:
Proportions of TS subjects achieving self-reported withdrawal bleeding (defined as spotting or bleeding episodes that occur at least for one day) during the treatment with Progynova or Oestrogel regimen | From enrollment to 19 months after the commencement of intervention (end of follow-up)
  Self-reported by patients through documentation in a personal diary
Median time to withdrawal bleeding (in days) | From enrollment to 19 months after the commencement of intervention (end of follow up)
  The exact number of days of the time from the commencement of intervention until the occurrence of the first withdrawal bleeding. The occurrence of the first withdrawal bleeding is self-reported by patients through documentation in a personal diary. Withdrawal bleeding is defined as the occurrence of at least spotting (defined as bloody discharge that requires not more than a panty liner) based on Zhang and colleagues' criteria (reference 36)
Serum Triglyceride levels (in mmol/L) | From enrollment to 19 months after the commencement of intervention (end of follow-up)
  Serum triglyceride level of the participant as reported by the laboratory based on the blood samples taken during the follow-ups at the PAG unit of HCTM.

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD IRFAN ABDUL JALAL, MBChB BAO, PhD, Study Chair — Universiti Kebangsaan Malaysia Medical Molecular Biology Institute (UMBI); ANI AMELIA ZAINUDDIN, MBBS, PhD, Principal Investigator — FACULTY OF MEDICINE, UNIVERSITI KEBANGSAAN MALAYSIA; NUR AZURAH ABDUL GHANI, MBBS, MMed (Obs and Gynae), Principal Investigator — National University of Malaysia
Locations (1):
- Hospital Canselor Tuanku Muhriz (HCTM), Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
The final and cleaned-up version of the trial dataset containing individual clinical-trial participant data (IPD) for all study variables will be deposited in a public repository such as the Harvard Dataverse data repository (available from: https://dataverse.harvard.edu/) to ensure the transparency of trial reporting and compliance with the clinicaltrials.gov data sharing policies. The preliminary trial results will first be uploaded into the clinicaltrials.gov registry within 6 months after the completion of the last patient visit for early dissemination of trial results.
  The final trial findings (including trial objectives, the design of the trial (including revisions), the statistical analysis plan (including amendments) and the originally planned measurements of efficacy and safety parameters) will then be published as presentations at scientific conferences and in a complete published manuscript, even if the trial has to be prematurely halted.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 01/11/2029 until 31/10/2039 (10 years)
Access Criteria: The general public and all researchers will have access to the IPD. The supporting information (full trial protocol and statistical analysis plan, informed consent form and case report form (CRF; English version) is available for download as separate study documents uploaded on this website.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2026-01-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT07041814/Prot_SAP_ICF_001.pdf